CLINICAL TRIAL: NCT02254850
Title: The Mesoglycan and Vascular Reactivity in the Metabolic Syndrome
Brief Title: Mesoglycan, Vascular Reactivity and Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ugo Oliviero, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Mesoglicano 29/13
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Metabolic Syndrome
Keywords: Mesoglycan; Metabolic Syndrome; Flow Mediated Dilation
MeSH Terms: conditions — Metabolic Syndrome | interventions — mesoglycan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesoglycan (Experimental): The Patients firstly underwent to intramuscular administration of 1 vial only, containing: Mesoglycan 30mg/ml and inactive ingredients: sodium chloride, chlorocresol, water for injections.
  Nextly the patients underwent to oral treatment with 1 capsule, administered bis in die for a period of 90 days, containing: Mesoglycan 50 mg and Inactive ingredients: lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate, gelatin, titanium dioxide, erythrosine.
  Patients also performed Flow Mediated Dilation (FMD).
  Interventions: Procedure: Flow Mediated Dilation; Drug: Mesoglycan
- Placebo (Placebo Comparator): The Patients firstly underwent to intramuscular administration only of 1 vial containing inactive ingredients: sodium chloride, chlorocresol, water for injections.
  Nextly the patients underwent to oral treatment with 1 capsule, administered bis in die for a period of 90 days, containing inactive ingredients: lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate, gelatin, titanium dioxide, erythrosine.
  Patients also performed Flow Mediated Dilation (FMD).
  Interventions: Procedure: Flow Mediated Dilation; Drug: Placebo

INTERVENTIONS:
Procedure: Flow Mediated Dilation — Patients performed FMD by an high-resolution ultrasound linear probe in a supine decubitus and conditioned room.The probe was placed on humeral artery and connected to a mechanically arm. Then were performed several measurement s of the internal diameter of the vessel (edge to edge distance), on the R wave of the ECG, and "software" calculated the average value.The post-ischemic vasodilation was induced using a sphygmomanometer placed on the forearm, distal to the elbow crease, kept inflated to 250 mmHg for 5 minutes. The flow rate was recorded immediately after the desufflation; the diameter of the brachial artery was measured several times after desufflation (for 60-90 seconds). Nextly, the FMD was calculated as the percentage difference between the maximum diameter of the post-ischemic reached and the mean diameter of the vessel.
  Other Names: FMD
Drug: Mesoglycan — The Patients firstly underwent to intramuscular administration of 1 vial only, containing: Mesoglycan 30mg/ml.
  Other Names: Mesoglycan Intramuscular injecion
  Arms: Mesoglycan
Drug: Mesoglycan — The patients underwent to oral treatment with 1 capsule, administered bis in die for a period of 90 days, containing: Mesoglycan 50 mg.
  Other Names: Mesoglycan Oral Treatment
  Arms: Mesoglycan
Drug: Placebo — The Patients firstly underwent to intramuscular administration only of 1 vial containing inactive ingredients: sodium chloride, chlorocresol, water for injections.
  Other Names: Placebo Intramuscular Injection
  Arms: Placebo
Drug: Placebo — The patients underwent to oral treatment with 1 capsule, administered bis in die for a period of 90 days, containing inactive ingredients: lactose monohydrate, corn starch, croscarmellose sodium, magnesium stearate, gelatin, titanium dioxide, erythrosine.
  Other Names: Placebo Oral Treatment
  Arms: Placebo

SUMMARY:
The purpose of the study was to characterize the action of mesoglycan on vascular endothelium through the non-invasive assessment of vascular reactivity humeral artery by comparing effects of mesoglycan on Flow Mediated Dilatation (FMD) of the humeral artery between a group of patients with metabolic syndrome assuming placebo and a group of patient with metabolic syndrome assuming mesoglycan; firstly after administration of the drug/placebo intramuscularly, and then, in a study of medium-term after oral intake of drug/placebo. The selection of patients with metabolic syndrome is related to the fact that this syndrome is associated with alterations in endothelial function and a high incidence of cardiovascular events. So it is a condition that offers the opportunity to explore the hypothesis that the mesoglycan may have a favorable effect on early vascular alterations that precede clinical events.

DETAILED DESCRIPTION:
The subjects were enrolled in a double blind randomized way, according to a 2: 1 ratio, to intramuscular treatment with mesoglycan or placebo. Patients performed the study of the Flow Mediated Dilation (FMD) according to the following scheme:

* FMD baseline
* FMD 2 hours after the administration of 2 vials of mesoglycan or placebo intramuscularly
* FMD 6 hours after intramuscular administration.

Nextly, both patients treated with mesoglycan vials and placebo vials continued therapy for assuming mesoglycan or placebo, per os, bis in die, for 90 days. At the end of this period of oral therapy (mesoglycan or placebo in a 2: 1 ratio), all patients performed FMD again. The patients who were taking any specific therapy (eg antihypertensive drugs) the Placebo was administered in addition to their standard therapy.

The vascular reactivity evaluation adopted was the Flow Mediated Dilatation (FMD). After a period of fasting and rest for at least 6 hours, the study of FMD was performed using a high-resolution ultrasound system, equipped with a 7.5 Megahertz linear probe under ECG monitoring. After a rest period of at least 10 minutes on a bed in supine decubitus in an air-conditioned room, the sensor was placed on humeral artery, 3-5 cm above the elbow, and held the same position during the examination through an arm mechanically connected. They were performing a number of longitudinal sections and measured the internal diameter of the vessel, defined as the distance between the top edge of the echo produced by the interface between the lumen and the anterior wall of the vessel and the top edge of the echo produced by the interface between the lumen and the rear wall of the vessel. The inner diameter of the vessel was measured several times, on the R wave of the ECG, and a pc "software" calculated the average value. The flow rate was measured with the sample volume placed in the center of the vase with a 60 ° angle between the ultrasound beam and the longitudinal axis of the vessel. The post-ischemic vasodilation was induced using a sphygmomanometer placed on the forearm, distal to the elbow crease, kept inflated to 250 mmHg for 5 minutes. The flow rate, always with a correction angle of 60 °, was recorded immediately after the desufflation; the diameter of the brachial artery, it was measured several times after desufflation (for 60-90 seconds). Nextly, the FMD was calculated as the percentage difference between the maximum diameter of the post-ischemic reached and the mean diameter of the base of the vessel.

ELIGIBILITY:
Inclusion Criteria:

3 or more of the following criteria of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III):

* Increased abdominal circumference ≥102 cm in man, ≥88 cm in women
* Triglycerides ≥150 mg / dL
* HDL-cholesterol <40 mg / dL in men, <50 mg / dL in women
* Systolic blood pressure> 130 mm Hg or diastolic blood pressure> 85 mm Hg
* Blood glucose> 100 mg / dL

Exclusion Criteria:

* Indication for cardiac surgery or surgeries performed by less than 3 months
* Under the age of 18 years
* Age greater than 65 years
* Inability to perform periodic inspections
* Presence of malignancy and serious heart diseases.
* Hemorrhagic diathesis and diseases.
* Hypersensitivity to mesoglycan, heparin and heparinoids.
* Type 1 diabetes and type 2
* Pregnancy and / or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Improvement of FMD | 90 days
  Verify if taken chronically mesoglycan 1 cp morning and evening for 90 days change compared to placebo vascular reactivity in subjects with metabolic syndrome (increased FMD in the treated group compared to baseline after 90 days of therapy) .

SECONDARY OUTCOMES:
Improvement of FMD | 2 and 6 hours
  Verify if the mesoglycan administered intramuscularly change the vascular reactivity compared to placebo in subjects with metabolic syndrome (increased FMD from baseline in 2 and 6 hours after intramuscular administration)

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Oliviero, MD, Principal Investigator — Federico II University-Dipartimento di Scienze Mediche Traslazionali
Locations (1):
- Ugo Oliviero, Via Pansini, 5, Napoli, Italy

REFERENCES:
- [Background] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Costa F; American Heart Association; National Heart, Lung, and Blood Institute. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute Scientific Statement. Circulation. 2005 Oct 25;112(17):2735-52. doi: 10.1161/CIRCULATIONAHA.105.169404. Epub 2005 Sep 12. No abstract available. PMID 16157765
- [Background] Reaven G. The metabolic syndrome or the insulin resistance syndrome? Different names, different concepts, and different goals. Endocrinol Metab Clin North Am. 2004 Jun;33(2):283-303. doi: 10.1016/j.ecl.2004.03.002. PMID 15158520
- [Background] Balkau B, Charles MA. Comment on the provisional report from the WHO consultation. European Group for the Study of Insulin Resistance (EGIR). Diabet Med. 1999 May;16(5):442-3. doi: 10.1046/j.1464-5491.1999.00059.x. No abstract available. PMID 10342346
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Ridker PM, Wilson PW, Grundy SM. Should C-reactive protein be added to metabolic syndrome and to assessment of global cardiovascular risk? Circulation. 2004 Jun 15;109(23):2818-25. doi: 10.1161/01.CIR.0000132467.45278.59. PMID 15197153
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Prieto D, Contreras C, Sanchez A. Endothelial dysfunction, obesity and insulin resistance. Curr Vasc Pharmacol. 2014 May;12(3):412-26. doi: 10.2174/1570161112666140423221008. PMID 24846231
- [Background] Anderson TJ. Nitric oxide, atherosclerosis and the clinical relevance of endothelial dysfunction. Heart Fail Rev. 2003 Jan;8(1):71-86. doi: 10.1023/a:1022199021949. PMID 12652161
- [Background] Forconi S, Battistini N, Guerrini M, Passero SG for the SIAM Group. A randomized, ASA-controlled trial of mesoglycan in secondary prevention after cerebral ischemic events. Cerebrovasc Dis 1995; 5:334-341.
- [Background] Orefice G, Brancaccio V, Coppola G et al. Comparative effects of mesoglycan and ticlopidine treatment on some coagulative parameters in patients with previous ischemic stroke: results of a randomized controlled trial. Current Therapeutic Research 2002; 63:337-343.
- [Background] Nenci GG, Gresele P, Ferrari G, Santoro L, Gianese F; Mesoglycan Intermittent Claudication Group. Treatment of intermittent claudication with mesoglycan--a placebo-controlled, double-blind study. Thromb Haemost. 2001 Nov;86(5):1181-7. PMID 11816704
- [Background] Charakida M, Masi S, Luscher TF, Kastelein JJ, Deanfield JE. Assessment of atherosclerosis: the role of flow-mediated dilatation. Eur Heart J. 2010 Dec;31(23):2854-61. doi: 10.1093/eurheartj/ehq340. Epub 2010 Sep 23. PMID 20864485
- [Background] Tufano A, Arturo C, Cimino E, Di Minno MN, Di Capua M, Cerbone AM, Di Minno G. Mesoglycan: clinical evidences for use in vascular diseases. Int J Vasc Med. 2010;2010:390643. doi: 10.1155/2010/390643. Epub 2010 Aug 31. PMID 21152191
- [Background] Juhan-Vague I, Morange PE, Alessi MC. The insulin resistance syndrome: implications for thrombosis and cardiovascular disease. Pathophysiol Haemost Thromb. 2002 Sep-Dec;32(5-6):269-73. doi: 10.1159/000073579. PMID 13679655